CLINICAL TRIAL: NCT05401487
Title: Multicentre Study: Adherence to the Severe Trauma Patients Pathway in PACA Region
Acronym: FILTRAUMA-PACA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-CHITS-013
Record Dates: First submitted 2022-05-20; First posted 2022-06-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Trauma
Keywords: severe trauma; PACA ORU recommendations; golden hour; emergency rapid response unit; hospital care; prognosis
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patient with a severe trauma requiring SMUR activation: Trauma defined by appearance of lesions following a fall, a road accident, a burn or the penetration of a foreign body and regulated by one of the SAMU PACA region centres (84, 83, 13, 04)
  Interventions: Other: Pre-hospital and hospital care

INTERVENTIONS:
Other: Pre-hospital and hospital care — Pre-hospital care not exceeding 60 min and a whole body CT scan within 45 min for patients categorized as unstable or critical by the pre-hospital doctor and 90 minutes for patients deemed potentially serious.

SUMMARY:
Trauma patient management concerns more than 140,000 patients per year in France. PACA Regional Emergency Observatory (ORU) has issued recommendations to optimize the management of these trauma patients from pre-hospital phase to hospitalization first hours. Ideally, pre-hospital care should not exceed 60 minutes, from accident (first call to the SAMU) to trauma center arrival: the "golden hour" concept. Patients presenting at least one of the Vittel criteria are considered as severely traumatized and are classified according to 3 states of seriousness: unstable, critical and potentially serious. They are referred to trauma centers whose classification is based on their technical facilities, ranging from level 1 (maximum technical facilities) to level 3 (minimum technical facilities). Patients are referred according to their severity, distance from accident site, referral center and availability of each site. Initial hospital management recommends a whole body CT scan within 45 minutes for patients categorized as unstable or critical by pre-hospital doctor and 90 minutes for patients deemed potentially serious.

FILTRAUMA PACA study will analyze the impact of the different management sequences of severe trauma patients based on reliable temporal data because it is automatically incremented in databases and will seek to find a correlation with patient outcome (survival at 24 hours and 28 days).

The main hypothesis tested is that PACA ORU recommended delay respect during trauma patient initial management is correlated with vital prognosis in short (24 hours) and medium terms (28 days).

DETAILED DESCRIPTION:
Trauma patient management concerns more than 140,000 patients per year in France. Grenoble region was the first one to organize its trauma network around trauma centers ranked by levels (from level 1, the most complete technical platform, to level 3). PACA Regional Health Agency (ARS) set up its dedicated line for severe trauma patients in 2014 based on a regional multi-professional group recommendations, the PACA Regional Emergency Observatory (ORU), in order to optimize the management of these trauma patients from pre-hospital phase to hospitalization first hours (recommendations available online: https://ies-sud.fr/bonnes-pratiques/).

This network suggests a care pathway setting objectives at each stage with operating requirements. Ideally, pre-hospital care should not exceed 60 minutes, from accident (first call to the SAMU) to trauma center arrival: the "golden hour" concept. Patients presenting at least one of the Vittel criteria are considered as severely traumatized and are classified according to 3 states of seriousness: unstable, critical and potentially serious. They are referred to trauma centers whose classification is based on their technical facilities, ranging from level 1 (maximum technical facilities) to level 3 (minimum technical facilities). In PACA region, level 1 technical platforms are North Hospital and Timone Hospital (AP-HM, Marseille, 13) and Sainte Anne Hospital (Toulon, 83). Levels 2 are Sainte Musse Hospital (Toulon, 83), Saint Joseph Hospital (Marseille, 13) and Avignon Hospital (84) and levels 3 correspond to all other hospitals in the region. Patients are referred according to their severity, distance from accident site, referral center and availability of each site. Initial hospital management recommends a whole body CT scan within 45 minutes for patients categorized as unstable or critical by the pre-hospital doctor and 90 minutes for patients deemed potentially serious.

FILTRAUMA PACA study will analyze the impact of the different management sequences of severe trauma patients based on reliable temporal data because it is automatically incremented in databases and will seek to find a correlation with patient outcome (survival at 24 hours and 28 days). The main hypothesis tested is that PACA ORU recommended delay respect during trauma patient initial management is correlated with vital prognosis in short (24 hours) and medium terms (28 days).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any patient with a severe trauma requiring SMUR activation. Trauma defined by the appearance of a lesion following a fall, a road accident, a burn or the penetration of a foreign body and regulated by one of the PACA region SAMU centres (84, 83, 13, 04)

Exclusion Criteria:

* Opposition of the patient, family member or trusted person
* Patient under legal protection (guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with a severe trauma requiring SMUR activation
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
To evaluate whether compliance with the "golden hour", pre-hospital delay recommended by PACA ORU, influences severe trauma patient vital status. | 24 hours
  Pre-hospital management duration (from the call to the SAMU to arrival at trauma centres) will be derived according to PACA ORU recommendation (time inferior or superior to 1 hour), and will then be related to patient's vital status at 24 hours.

SECONDARY OUTCOMES:
To evaluate whether adherence to ORU PACA recommendations in terms of pre-hospital management delays influences severe trauma patient vital status at day 28 | 28 days
  Pre-hospital management duration (from the call to the SAMU to arrival at trauma centres) will be derived according to PACA ORU recommendation (inferior or superior 1 hour), and will then be related to patient's vital status at day 28.
To assess whether transport by suitable vehicle to appropriate health facility recommended by the ORU PACA influences the vital status of severe trauma patients. | 28 days
  The influence of adherence to ORU PACA recommendations on severe trauma patient vital status (at 24 hours and 28 days after trauma) will be evaluated according to transport by suitable vehicle to appropriate health facility
To assess whether accident categorization and assessment transfer to the SAMU recommended by the ORU PACA influences the vital status of severe trauma patients. | 28 days
  The influence of adherence to ORU PACA recommendations on severe trauma patient vital status (at 24 hours and 28 days after trauma) will be evaluated according to accident categorization and assessment transfer to the SAMU
To assess whether management on accident scene recommended by the ORU PACA influences the vital status of severe trauma patients. | 28 days
  The influence of adherence to ORU PACA recommendations on severe trauma patient vital status (at 24 hours and 28 days after trauma) will be evaluated according to management on accident scene
To assess whether overall assessment of severity recommended by the ORU PACA influences the vital status of severe trauma patients. | 28 days
  The influence of adherence to ORU PACA recommendations on severe trauma patient vital status (at 24 hours and 28 days after trauma) will be evaluated according to Overall assessment of severity.
To assess whether time required to perform a whole body CT scan recommended by the ORU PACA influences the vital status of severe trauma patients. | 28 days
  The influence of adherence to ORU PACA recommendations on severe trauma patient vital status (at 24 hours and 28 days after trauma) will be evaluated according to time required to perform a whole body CT scan.
To analyze risk factors for non-adherence to recommendations | 28 days
  The risk factors for non-adherence to recommendations will be identified through primary and first secondary outcome criteria analysis. They will then be described (structural, patient-related).
To analyze errors in referring severe trauma patients to an appropriate care facility | 28 days
  Identification and analysis of the reasons for mis-referrals of severe trauma patients to an approved care facility.

CONTACTS AND LOCATIONS:
Overall Officials: Marc FOURNIER, MD, PhD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (3):
- France (3):
  - Centre Hospitalier de Digne les Bains, Digne-les-Bains, Alpes-de-Haute-Provence
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var
  - Centre Hospitalier d'Avignon Henri Duffaut, Avignon, Vaucluse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bege T, Pauly V, Orleans V, Boyer L, Leone M. Epidemiology of trauma in France: mortality and risk factors based on a national medico-administrative database. Anaesth Crit Care Pain Med. 2019 Oct;38(5):461-468. doi: 10.1016/j.accpm.2019.02.007. Epub 2019 Feb 23. PMID 30807878
- [Background] Gauss T, Balandraud P, Frandon J, Abba J, Ageron FX, Albaladejo P, Arvieux C, Barbois S, Bijok B, Bobbia X, Charbit J, Cook F, David JS, Maurice GS, Duranteau J, Garrigue D, Gay E, Geeraerts T, Ghelfi J, Hamada S, Harrois A, Kobeiter H, Leone M, Levrat A, Mirek S, Nadji A, Paugam-Burtz C, Payen JF, Perbet S, Pirracchio R, Plenier I, Pottecher J, Rigal S, Riou B, Savary D, Secheresse T, Tazarourte K, Thony F, Tonetti J, Tresallet C, Wey PF, Picard J, Bouzat P; Groupe d'interet en traumatologie grave (GITE). Strategic proposal for a national trauma system in France. Anaesth Crit Care Pain Med. 2019 Apr;38(2):121-130. doi: 10.1016/j.accpm.2018.05.005. Epub 2018 May 29. PMID 29857186
- [Background] Harmsen AM, Giannakopoulos GF, Moerbeek PR, Jansma EP, Bonjer HJ, Bloemers FW. The influence of prehospital time on trauma patients outcome: a systematic review. Injury. 2015 Apr;46(4):602-9. doi: 10.1016/j.injury.2015.01.008. Epub 2015 Jan 16. PMID 25627482
- [Background] Ashburn NP, Hendley NW, Angi RM, Starnes AB, Nelson RD, McGinnis HD, Winslow JE, Cline DM, Hiestand BC, Stopyra JP. Prehospital Trauma Scene and Transport Times for Pediatric and Adult Patients. West J Emerg Med. 2020 Feb 21;21(2):455-462. doi: 10.5811/westjem.2019.11.44597. PMID 32191204
- [Background] Mann NC, Mullins RJ, MacKenzie EJ, Jurkovich GJ, Mock CN. Systematic review of published evidence regarding trauma system effectiveness. J Trauma. 1999 Sep;47(3 Suppl):S25-33. doi: 10.1097/00005373-199909001-00007. PMID 10496607